CLINICAL TRIAL: NCT01854229
Title: A Prospective, Non-randomized, Open-label, Multicenter Study to Evaluate the Long-term Safety of the Prometra Programmable Pump System
Brief Title: Prometra Post-Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flowonix Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAS-01
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain; Cancer Pain; Intractable Pain; Back Pain
Keywords: Morphine; Implantable Infusion Pumps; Intrathecal Pump
MeSH Terms: conditions — Chronic Pain; Cancer Pain; Pain, Intractable; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prospective pump candidates (Active Comparator): New candidates who will receive the Prometra Programmable Intrathecal Infusion Pump
  Interventions: Device: Prometra Programmable Intrathecal Infusion Pump
- Previous IDE study subjects continuing with the therapy (Active Comparator): Patients who were part of the previous IDE study, still have an active Prometra Programmable Intrathecal Infusion Pump, and are willing to continue in a study protocol.
  Interventions: Device: Prometra Programmable Intrathecal Infusion Pump

INTERVENTIONS:
Device: Prometra Programmable Intrathecal Infusion Pump — There are two enrollment groups (arms). One is for new patients who are going to have a Prometra Pump implanted. The other arm is for patients who were part of the IDE study prior to FDA approval of the pump, and are willing to continue to be followed as part of a study.
  Other Names: Flowonix pump

SUMMARY:
The Prometra Pump is approved by the FDA for use in the United States. The purpose of this study is to collect long-term safety data on the Prometra Pump.

DETAILED DESCRIPTION:
This study is proposed under part of the post-Premarket Approval (PMA) requirements. This study is a prospective, non-randomized, open-label, multicenter study. It will be performed at 10-30 centers in the US and enroll a maximum of 400 subjects. Subjects will be followed for a total of five years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient meets at least one of the following:

   * is suffering from malignant pain (i.e., cancer pain)
   * has chronic, non-malignant pain
   * subject was enrolled in PUMP I or PUMP II study and chooses to participate in this Post-Approval study
   * Patient with an existing implantable pump for pain therapy that requires replacement
2. Patient is at least 22 years of age.
3. Investigator considers the patient to be able and willing to fulfill all study requirements.
4. Patient has provided written informed consent to participate in the study.

Exclusion Criteria:

1. Patient meets any of the contraindications for use of the Prometra System
2. Patient has a prior history of granuloma formation, or is receiving treatment for a suspected granuloma.
3. Patient is pregnant or breast-feeding or is of child-bearing potential and not employing effective birth control.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Rate of granuloma formation | Five years
  The primary hypothesis is that the 5-year rate of patients with granuloma formation will be noninferior to that in the literature. The literature rate was found to be approximately 3% and the noninferiority margin will be three percentage points.

SECONDARY OUTCOMES:
Pump failure | Five years
  Tabulation of pump failures, including time to occurrence and type
Pump battery life | Five years
  Tabulation of occurences of premature pump battery depletions

OTHER OUTCOMES:
Device-related adverse events | Five years
  Tabulation of device-related adverse events
Device-related serious adverse events | Five years
  Tabulation of device-related serious adverse events
Rate of granuloma formation by race and ethnicity | Five years
  The effect of race and ethnicity on granuloma formation
Granuloma formation by drug type | Five years
  The effect of alternative drugs on granuloma formation

CONTACTS AND LOCATIONS:
Overall Officials: Cory Brantley, Study Director — Flowonix Medical
Locations (26):
- United States (26):
  - Perlman Clinic, La Jolla, California
  - Pacific Pain Physicians, Santa Barbara, California
  - Evolve Restorative Center, Santa Barbara, California
  - Summit Pain Alliance, Santa Rosa, California
  - BioHealth Pain Management, Torrance, California
  - Interventional Pain Management, Daytona Beach, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Palm Beach Pain Management, Lake Worth, Florida
  - Pain Institute of Tampa, Tampa, Florida
  - Global Scientific Innovations, Evansville, Indiana
  - Summit Pain Management, Fort Wayne, Indiana
  - Summit Research Institute, Fort Wayne, Indiana
  - Interventional Pain Management Specialists, Overland Park, Kansas
  - Bluegrass Pain Consultants, Louisville, Kentucky
  - Kentuckiana Pain Specialists, Louisville, Kentucky
  - Neuroscience and Pain Institute, Covington, Louisiana
  - Integrated Pain and Neuroscience, New Orleans, Louisiana
  - Jackson Anesthesia Pain Center, Jackson, Mississippi
  - Triumph Medical, Asheville, North Carolina
  - Integrated Pain Solutions, Columbus, Ohio
  - Pain Management Institute, Wooster, Ohio
  - Neurospine Institute, Eugene, Oregon
  - Pain Care of Oregon, Medford, Oregon
  - Fox Chase Pain Management Associates, Trevose, Pennsylvania
  - Space City Pain Specialists, Webster, Texas
  - Nexus Pain Care, Provo, Utah

REFERENCES:
- [Background] Rauck R, Deer T, Rosen S, Padda G, Barsa J, Dunbar E, Dwarakanath G. Long-term follow-up of a novel implantable programmable infusion pump. Neuromodulation. 2013 Mar-Apr;16(2):163-7. doi: 10.1111/j.1525-1403.2012.00515.x. Epub 2012 Oct 11. PMID 23057877
- See also: American Academy of Pain Medicine — http://www.painmed.org/
- See also: North American Neuromodulation Society — http://www.neuromodulation.org/
- See also: American Society of Regional Anesthesia and Pain Medicine — http://www.asra.com/
- See also: World Institute of Pain — https://www.worldinstituteofpain.org